CLINICAL TRIAL: NCT00843726
Title: A Phase II Randomized Study of 2 Stereotactic Body Radiation Therapy (SBRT) Regimens for Medically Inoperable Patients With Node Negative, Peripheral Non-Small Cell Lung Cancer
Brief Title: Radiation Therapy in Treating Patients With Stage I or Stage II Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 124407; I 124407 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients undergo 1 high-dose fraction of stereotactic body radiotherapy (SBRT).
  Interventions: Radiation: Arm 1 stereotactic body radiation therapy
- Arm II (Experimental): Patients undergo 3 high-dose fractions (approximately 1 week apart) of SBRT.
  Interventions: Radiation: Arm II stereotactic body radiation therapy

INTERVENTIONS:
Radiation: Arm 1 stereotactic body radiation therapy — Patients undergo 1 high-dose fraction
  Arms: Arm I
Radiation: Arm II stereotactic body radiation therapy — Patients undergo 3 high-dose fractions
  Arms: Arm II

SUMMARY:
RATIONALE: Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue. It is not yet known which regimen of radiation therapy is more effective in treating patients with non-small cell lung cancer.

PURPOSE: This randomized phase II trial is studying the side effects of two radiation therapy regimens and to see how well they work in treating patients with stage I or stage II non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the incidence of toxicity with two established stereotactic body radiotherapy (SBRT) regimens in patients with node-negative, peripheral stage I or II non-small cell lung cancer.

Secondary

* To compare quality of life, patterns of failure, disease-free survival, and overall survival of these patients after treatment with one of two established SBRT regimens.
* To correlate outcomes and toxicities with imaging and patient and tumor biomarkers.

OUTLINE: Patients are stratified according to Karnofsky performance status and treatment center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo 1 high-dose fraction of stereotactic body radiotherapy (SBRT).
* Arm II: Patients undergo 3 high-dose fractions (approximately 1 week apart) of SBRT.

Quality of life is assessed periodically by the EORTC QLQ-C30 and -LC13 questionnaires

Blood and tissue samples may be collected periodically and examined for biomarkers via ELISA and immunoblotting.

After completion of study treatment, patients are followed for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer
* T1-T2, N0 disease measuring ≤ 5 cm( T3 tumor based on chest wall involvement is Excluded)
* Surgically resectable primary disease, however patient evaluated by thoracic oncologist and deemed medically inoperable OR patient refuses surgical resection
* Age >= 18

Exclusion Criteria:

* Prior thoracic radiation therapy
* T2 or T3 tumor greater than 5 cm or T3 tumor based on chest wall involvement
* Node positive or metastatic disease
* Tumor location within the zone of the proximal bronchial tree. The proximal bronchial tree is defined as the carina, right and left main bronchi, right and left upper lobe bronchi, bronchus intermedius, right middle lobe bronchus, lingular bronchus, and right and left lower lobe bronchi. The zone of the proximal bronchial tree is defined as a volume 2cm in all directions around the proximal bronchial tree.
* No other conditions deemed by the PI or associates to make the patient ineligible for protocol investigations, procedures, and high-dose external beam radiotherapy (e.g., unable to lie still and breathe reproducibly)
* Pregnant or unwilling to use adequate contraception

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2008-09-12 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anurag K. Singh, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (3):
- United States (3):
  - Roswell Park Cancer Institute, Buffalo, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Cleveland Clinic, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 High-dose Fraction SBRT: Patients undergo 1 high-dose fraction of stereotactic body radiotherapy (SBRT).
  stereotactic body radiation therapy: Patients undergo 1 high-dose fraction
- 3 High-dose Fractions SBRT: Patients undergo 3 high-dose fractions (approximately 1 week apart) of SBRT.
  stereotactic body radiation therapy: Patients undergo 3 high-dose fractions
Period: Overall Study
Arm/Group | 1 High-dose Fraction SBRT | 3 High-dose Fractions SBRT
Started | 49 | 49
Completed | 48 | 48
Not Completed | 1 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 High-dose Fraction SBRT | 3 High-dose Fractions SBRT | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 2 | 7 | 9
  >=65 years | 45 | 40 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.5 (7.5) | 74.5 (8.0) | 75.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 50
  Male | 22 | 26 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 41 | 43 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Incidence of AE Grade 3 or Higher Toxicity
Description: Count of patients experiencing at least one grade 3 or higher adverse event. The Common Terminology Criteria for Adverse Events (CTCAE) v3.0 is used for assessing the adverse events. High grades AEs are considered worse.
Time Frame: 1year
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Groups:
- I High-dose Fraction SBRT: Patients undergo 1 high-dose fraction of stereotactic body radiotherapy (SBRT).
  stereotactic body radiation therapy: Patients undergo 1 high-dose fraction
Arm/Group | I High-dose Fraction SBRT | 3 High-dose Fractions SBRT
Number analyzed (Participants) | 49 | 49
Participants | 24 | 26

2. Primary Outcome: Overall Survival
Description: Median overall survival
Time Frame: 5 years
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1 High-dose Fraction SBRT | 3 High-dose Fractions SBRT
Number analyzed (Participants) | 49 | 49
months | 39.0 [27.2 to 51.9] | 38.3 [21.1 to 49.0]

3. Primary Outcome: Correlation Between Blood and Serum Markers and Survival and Toxicity
Time Frame: 4 years
Population: Data was not collected for this outcome
Arm/Group | 1 High-dose Fraction SBRT | 3 High-dose Fractions SBRT
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline, weekly until 30 day follow-up.
Arm/Group | 1 High-dose Fraction SBRT | 3 High-dose Fractions SBRT
All-Cause Mortality (participants affected / at risk) | 33/49 | 29/49
Serious Adverse Events (participants affected / at risk) | 2/49 | 5/49
Other Adverse Events (participants affected / at risk) | 38/49 | 36/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 High-dose Fraction SBRT (N=49) | 3 High-dose Fractions SBRT (N=49)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 High-dose Fraction SBRT (N=49) | 3 High-dose Fractions SBRT (N=49)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 3 (5)
Chills (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 18 (21) | 21 (22)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (4) | 3 (3)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 11 (12)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT00843726/Prot_SAP_000.pdf